CLINICAL TRIAL: NCT00084305
Title: Analysis of Specimens From Individuals With Pulmonary Fibrosis
Status: Active, not recruiting | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040211; 04-HG-0211
Record Dates: First submitted 2004-06-09; First posted 2004-06-10 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-06

CONDITIONS: Pulmonary Fibrosis; Healthy Volunteers; Hermansky-Pudlak Syndrome (HPS)
Keywords: Bronchoscopy; Pulmonary Fibrosis; Lung Biopsy (Clinically-Indicated); Natural History
MeSH Terms: conditions — Pulmonary Fibrosis; Hermanski-Pudlak Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Family: Family members of patients with pulmonary fibrosis
- Healthy Volunteers: Healthy Volunteers
- Pulmonary Fibrosis: Patients with pulmonary fibrosis

SUMMARY:
The etiology of pulmonary fibrosis is unknown. Analyses of blood, genomic DNA, and specimens procured by bronchoscopy, lung biopsy, lung transplantation, clinically-indicated extra-pulmonary biopsies, or post-mortem examination from individuals with this disorder may contribute to our understanding of the pathogenic mechanisms of pulmonary fibrosis. The purpose of this protocol is to procure and analyze blood, genomic DNA, and specimens by bronchoscopy, lung biopsy, lung transplantation, extra-pulmonary biopsies, or post-mortem examination from subjects with pulmonary fibrosis. In addition, blood, genomic DNA, clinically-indicated extra-pulmonary biopsies, as well as bronchoscopy and post-mortem examination specimens may be procured and analyzed from relatives of subjects with hereditary forms of pulmonary fibrosis; blood, genomic DNA, and bronchoscopy specimens may be procured from healthy research volunteers....

DETAILED DESCRIPTION:
The etiology of pulmonary fibrosis is unknown. Analyses of blood, genomic DNA, and specimens procured by bronchoscopy, lung biopsy, lung transplantation, clinically-indicated extra-pulmonary biopsies, or post-mortem examination from individuals with this disorder may contribute to our understanding of the pathogenic mechanisms of pulmonary fibrosis. The purpose of this protocol is to procure and analyze blood, genomic DNA, and specimens by bronchoscopy, lung biopsy, lung transplantation, extra-pulmonary biopsies, or post-mortem examination from subjects with pulmonary fibrosis. In addition, blood, genomic DNA, clinically-indicated extra-pulmonary biopsies, as well as bronchoscopy and post-mortem examination specimens may be procured and analyzed from relatives of subjects with hereditary forms of pulmonary fibrosis; blood, genomic DNA, and bronchoscopy specimens may be procured from healthy research volunteers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who are 18 years of age or older with any of the following:

* Idiopathic pulmonary fibrosis [defined by the American Thoracic Society/European Respiratory Society guidelines],
* Familial pulmonary fibrosis [defined as idiopathic pulmonary fibrosis in two or more first-degree relatives],
* Relatives of patients with hereditary pulmonary fibrosis,
* Hermansky-Pudlak syndrome (diagnosed by paucity or deficiency of platelet dense bodies on whole mount electron microscopy or by genetic testing),
* Pulmonary fibrosis associated with collagen vascular diseases or autoinflammatory disorders,
* Pulmonary fibrosis post-COVID-19 [i.e., pulmonary fibrosis in an individual recovering from SARS-CoV-2 infection], or
* Healthy research volunteers by history and indicated tests (individuals without history of chronic pulmonary disorder, collagen vascular disease, or bleeding disorder).

EXCLUSION CRITERIA:

Individuals with any of the following:

* Significant inhalational exposure to fibrogenic fibers or dusts or exposure to drugs associated with pulmonary fibrosis,
* Uncontrolled ischemic heart disease,
* Uncorrectable bleeding diathesis,
* Pregnancy or lactation (excluded due to exposure of unnecessary risks), or
* Inability to give informed consent (excluded due to exposure of unnecessary risks).

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary fibrosis@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2004-06-09 (Actual)

PRIMARY OUTCOMES:
Procure and analyze | Ongoing
  The objectives and specific aims of this protocol are to procure and analyze blood and cell/tissue specimens from individuals with pulmonary fibrosis, relatives of subjects with familial pulmonary fibrosis, and healthy research volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Introne, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Han CG, O'Brien KJ, Coon LM, Majerus JA, Huryn LA, Haroutunian SG, Moka N, Introne WJ, Macnamara E, Gahl WA, Malicdan MCV, Chen D, Krishnan K, Gochuico BR. Severe bleeding with subclinical oculocutaneous albinism in a patient with a novel HPS6 missense variant. Am J Med Genet A. 2018 Dec;176(12):2819-2823. doi: 10.1002/ajmg.a.40514. Epub 2018 Oct 4. PMID 30369044
- [Derived] El-Chemaly S, Cheung F, Kotliarov Y, O'Brien KJ, Gahl WA, Chen J, Perl SY, Biancotto A, Gochuico BR. The Immunome in Two Inherited Forms of Pulmonary Fibrosis. Front Immunol. 2018 Jan 31;9:76. doi: 10.3389/fimmu.2018.00076. eCollection 2018. PMID 29445374
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-HG-0211.html